CLINICAL TRIAL: NCT01928732
Title: CSP #591 - CERV-PTSD: Comparative Effectiveness Research in Veterans With PTSD
Brief Title: Comparative Effectiveness Research in Veterans With PTSD
Acronym: CERV-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 591
Record Dates: First submitted 2013-08-16; First posted 2013-08-27 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPT (Active Comparator): Cognitive Processing Therapy (CPT) - a type of cognitive therapy for treating PTSD.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)
- PE (Active Comparator): Prolonged Exposure (PE) - a type of exposure therapy for treating PTSD.
  Interventions: Behavioral: Prolonged Exposure (PE)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — CPT consists of cognitive therapy and a written trauma narrative. Patients are taught to challenge their beliefs through Socratic questioning and the use of daily worksheets. The initial focus is on beliefs such as denial and self-blame, and then shifts to overgeneralized beliefs about self and the world. Patients process their trauma directly by writing a narrative of their traumatic event(s) that they read to themselves and to therapists. The typical protocol consists of 12 1-hr sessions. In this study, the 12-session protocol will be followed, but participants who improve more rapidly may finish in 10 sessions and those who improve more slowly may receive up to 2 additional sessions to continue working on stuck points with challenging beliefs worksheets.
  Arms: CPT
Behavioral: Prolonged Exposure (PE) — PE is a manualized, 90-minute, 8-15 week treatment program based on emotional processing theory, which posits that anxiety disorders, including PTSD, reflect pathological fear structures in which emotional and cognitive associations among different elements do not accurately represent reality and renders the individual dysfunctional and distressed. PE is designed to correct erroneous connections in the targeted memory structure. PTSD sufferers typically experience two key pathological emotional response sets and related cognitions: "The world is an utterly dangerous place," and "I am completely incompetent and unable to cope with stress." In this study, the 12-session protocol will be followed, but participants improve more rapidly may finish in 10 sessions and those who improve more slowly may have up to 2 additional sessions to continue working on exposure.
  Arms: PE

SUMMARY:
VA Cooperative Study CSP #591 is designed to compare the effectiveness of two types of psychotherapy, Prolonged Exposure (PE) and Cognitive Processing Therapy (CPT), for treating posttraumatic stress disorder (PTSD) in male and female Veterans. Despite solid evidence that both treatments are effective in Veterans and non-Veterans, there is a lack of evidence about the effectiveness of these treatments compared with one another.

The sample will include 900 male and female Veterans with PTSD due to any traumatic military event. Veterans who are eligible and agree to participate in the study will be randomly assigned (by chance) to receive Prolonged Exposure or Cognitive Processing Therapy. The standard "dose" of treatment is 12 weekly sessions but Veterans who improve more rapidly may finish in fewer sessions and Veterans who improve more slowly may have additional sessions. The primary outcome is improvement in PTSD symptoms after treatment. The outcome will be measured at regular follow-up visits that will occur at the middle and at the end of treatment and then 3 and 6 months later. The investigators will measure other outcomes, including additional mental health problems, functioning, quality of life, and use of treatments for mental and physical problems. The investigators also will measure Veterans' treatment preference and examine whether Veterans who get the treatment they prefer do better than Veterans who get the less-preferred treatment.

As a large multi-site trial with men and women, CSP #591 is designed to provide conclusive information about whether one treatment is better than the other, overall and for different types of patients-for example, men vs. women, combat Veterans vs. Veterans who experienced military sexual trauma, and older vs. younger Veterans. Regardless of the outcome, patients will have more information to help them make an informed decisions about which treatment to choose and VA will have stronger evidence to help make care Veteran-centered.

DETAILED DESCRIPTION:
VA Cooperative Study CSP #591 is designed to compare the effectiveness of Prolonged Exposure (PE) and Cognitive Processing Therapy (CPT) for treating posttraumatic stress disorder (PTSD) in male and female Veterans. PTSD is a serious and prevalent condition in Veterans, affecting just under 9% of VA patients in Fiscal Year 2011 (FY11). Since 2005, the number of VA patients with PTSD has increased 14.8% annually, due not only to new Veterans but also to increased numbers of Vietnam Veterans who are seeking care. In FY11, PTSD was the 3rd most common service-connected disability in VA.

Despite solid evidence that Prolonged Exposure and Cognitive Processing Therapy are effective treatments for PTSD in Veterans and non-Veterans, there is insufficient evidence about the effectiveness of these treatments relative to one another. The only study to compare the treatments, a single-site trial in non-Veteran female rape survivors, failed to find a difference, but the study was not adequately powered to compare two such effective treatments. Other data are similarly inconclusive. CSP #591 would break new ground as the first large-scale comparative effectiveness trial of treatment for PTSD and the first study to provide definitive information about how effective treatments for PTSD compare with one another.

The study will be a prospective randomized clinical trial with blinded assessment. The population will be male and female Veterans with PTSD due to any traumatic military event. Patients who are eligible and agree to participate in the study will be randomly assigned in a 1:1 ratio to receive Prolonged Exposure or Cognitive Processing Therapy. The investigators propose to administer 12 weekly sessions of each treatment as a standard "dose" but to allow participants who improve more rapidly to finish in 10 or 11 sessions and participants who have not attained adequate improvement by session 12 to have up to 2 additional sessions.

The primary outcome is improvement in PTSD symptom severity as measured by change on the Clinician-Administered PTSD Scale after treatment. The outcome measure will be determined from regular follow-up visits of the patients, which will occur at the middle and at the end of treatment and then 3 and 6 months later. Secondary outcomes include other measures of PTSD, comorbid mental health problems, functioning, quality of life, and service utilization. The investigators also will measure participants' treatment preference and examine whether concordance between preference and allocation is associated with increased treatment effectiveness.

In order to detect a standardized mean difference in improvement in PTSD symptom severity of d = .25, a sample size of 900 randomized patients provides 90% power to detect a difference between arms using the linear mixed effects model with a two-sided = .05. Given the lack of conclusive findings to predict which treatment is better, the investigators propose to test a nondirectional hypothesis. Assuming 2.5 years of accrual and an enrollment of 26 participants per year at each site, the investigators would need 14.1 sites to enroll a total of 64 participants per site. The investigators propose to recruit 17 sites to guard against the possibility that some sites will not enroll the required number of participants.

VA has a vested interest in understanding the relative effectiveness of Prolonged Exposure and Cognitive Processing Therapy. Both treatments are recommended at the highest level in the Veterans Affairs (VA)/Department of Defense (DoD) PTSD Practice Guideline. VA is required to make these treatments available to Veterans seeking PTSD care. The treatments are being disseminated nationally across the VA system in order to enhance the availability of evidence-based treatments to Veterans with PTSD. VA also has developed a national PTSD Mentoring Program for PTSD Program Administrators to help them manage their clinics to permit the delivery of these treatments. Every facility has an evidence-based therapy coordinator as well to facilitate training in evidence-based psychotherapy.

As a large multi-site trial with men and women, CSP #591 would provide definitive information about the comparative effectiveness of Prolonged Exposure and Cognitive Processing Therapy and maximize the study's impact on the field. Because the treatments are based on differing theories about the development of PTSD, a demonstration that one treatment is superior to the other would further scientific exploration by challenging theoretical accounts of etiology and treatment. Regardless of which treatment is better, patients would have more information to help them make an informed decision about which treatment to choose and VA would have stronger evidence to help make care Veteran-centered.

ELIGIBILITY:
Inclusion Criteria:

Current PTSD and symptom severity of 25 or higher on the Clinician- Administered PTSD Scale (Weathers et al., 2013); agreement to not receive psychotherapy for PTSD during study treatment and allow digital recording of phone interviews and therapy; regular access to a telephone (or agreement to come to the VA for centrally conducted telephone interviews for participant who do not have telephone access). Medication for PTSD and other mental or physical conditions, psychotherapy for other problems, brief visits with an existing therapist, and self-help groups will be allowed.

Exclusion Criteria:

* substance dependence not in remission for at least 1 month;
* current psychotic symptoms and mania (including manic phase of bipolar disorder);
* significant current suicidal or homicidal ideation that includes a specific plan;
* or moderate to severe cognitive impairment defined as 1 SD below age-graded norms on the Montreal Cognitive Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 916 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula P Schnurr, PhD, Study Chair — White River Junction VA Medical Center, White River Junction, VT; Josef I Ruzek, PhD, Study Chair — VA Palo Alto Health Care System, Palo Alto, CA; Kathleen M Chard, PhD, Study Chair — Cincinnati VA Medical Center, Cincinnati, OH
Locations (18):
- United States (18):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnurr PP, Chard KM, Ruzek JI, Chow BK, Shih MC, Resick PA, Foa EB, Marx BP, Huang GD, Lu Y. Corrigendum to "Design of VA Cooperative Study #591: CERV-PTSD, Comparative Effectiveness Research in Veterans with PTSD" [Contemp. Clin. Trials 41 (2015) 75-84]. Contemp Clin Trials. 2019 May;80:61. doi: 10.1016/j.cct.2019.04.003. Epub 2019 Apr 5. No abstract available. PMID 30962124
- [Background] Schnurr PP, Chard KM, Ruzek JI, Chow BK, Shih MC, Resick PA, Foa EB, Marx BP, Huang GD, Lu Y. Design of VA Cooperative Study #591: CERV-PTSD, comparative effectiveness research in veterans with PTSD. Contemp Clin Trials. 2015 Mar;41:75-84. doi: 10.1016/j.cct.2014.11.017. Epub 2014 Nov 29. PMID 25457792
- [Result] Schnurr PP, Chard KM, Ruzek JI, Chow BK, Resick PA, Foa EB, Marx BP, Friedman MJ, Bovin MJ, Caudle KL, Castillo D, Curry KT, Hollifield M, Huang GD, Chee CL, Astin MC, Dickstein B, Renner K, Clancy CP, Collie C, Maieritsch K, Bailey S, Thompson K, Messina M, Franklin L, Lindley S, Kattar K, Luedtke B, Romesser J, McQuaid J, Sylvers P, Varkovitzky R, Davis L, MacVicar D, Shih MC. Comparison of Prolonged Exposure vs Cognitive Processing Therapy for Treatment of Posttraumatic Stress Disorder Among US Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2136921. doi: 10.1001/jamanetworkopen.2021.36921. PMID 35044471
- [Derived] Moshier SJ, Mahoney CT, Bovin MJ, Marx BP, Schnurr PP. Session-level effects of cognitive processing therapy and prolonged exposure on individual symptoms of posttraumatic stress disorder among U.S. veterans. J Consult Clin Psychol. 2024 Jul;92(7):422-431. doi: 10.1037/ccp0000880. Epub 2024 Mar 28. PMID 38546622

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral: Prolonged Exposure (PE): PE is a manualized, 90-minute, 8-15 week treatment program based on emotional processing theory, which posits that anxiety disorders, including PTSD, reflect pathological fear structures in which emotional and cognitive associations among different elements do not accurately represent reality and renders the individual dysfunctional and distressed. PE is designed to correct erroneous connections in the targeted memory structure. PTSD sufferers typically experience two key pathological emotional response sets and related cognitions: "The world is an utterly dangerous place," and "I am completely incompetent and unable to cope with stress." In this study, the 12-session protocol will be followed, but participants improve more rapidly may finish in 10 sessions and those who improve more slowly may have up to 2 additional sessions to continue working on exposure.
- Behavioral: Cognitive Processing Therapy (CPT): CPT consists of cognitive therapy and a written trauma narrative. Patients are taught to challenge their beliefs through Socratic questioning and the use of daily worksheets. The initial focus is on beliefs such as denial and self-blame, and then shifts to overgeneralized beliefs about self and the world. Patients process their trauma directly by writing a narrative of their traumatic event(s) that they read to themselves and to therapists. The typical protocol consists of 12 1-hr sessions. In this study, the 12-session protocol will be followed, but participants who improve more rapidly may finish in 10 sessions and those who improve more slowly may receive up to 2 additional sessions to continue working on stuck points with challenging beliefs worksheets.
Period: Overall Study
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Started | 455 | 461
Completed | 326 | 334
Not Completed | 129 | 127

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT) | Total
Number analyzed (Participants) | 455 | 461 | 916
Age, Continuous [Mean (Full Range); unit: years] | 45.5 [44.3 to 46.8] | 44.9 [43.7 to 46.1] | 45.2 [44.3 to 46.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 186
  Male | 361 | 369 | 730
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could select multiple categories for "Race."
  Participants
    White | 301 | 289 | 590
    Black | 119 | 130 | 249
    American Indian/Alaskan Native | 18 | 15 | 33
    Asian | 14 | 11 | 25
    Native Hawaiian/Pacific Islander | 7 | 10 | 17
    Other | 21 | 25 | 46
Service Era [Count of Participants; unit: Participants] — Service era was coded by including any Vietnam, Gulf, or OEF/OIF/OND veteran in their respective categories (including if they served in more than one era, e.g., Vietnam and Gulf). If a veteran did not serve in Vietnam, Gulf, or OEF/OIF/OND, they were coded as "Other."
  Participants
    Vietnam | 82 | 77 | 159
    Gulf War | 85 | 87 | 172
    OEF/OIF/OND | 260 | 270 | 530
    Other | 66 | 59 | 125
Post-high school education [Count of Participants; unit: Participants] | 216 | 192 | 408
Unemployed [Count of Participants; unit: Participants] | 271 | 263 | 534
Married/cohabitating [Count of Participants; unit: Participants] | 246 | 237 | 483
Ethnicity: Spanish, Hispanic or Latino [Count of Participants; unit: Participants] | 67 | 72 | 139
Positive VA Military Sexual Trauma Screen [Count of Participants; unit: Participants] | 134 | 133 | 267
Positive VA Traumatic Brain Injury Screen [Count of Participants; unit: Participants] | 294 | 281 | 575
Lifetime trauma exposure: Number of event types (of 17) [Mean (Full Range); unit: number of event types] | 7.7 [7.4 to 7.9] | 7.4 [7.2 to 7.7] | 7.54 [7.4 to 7.7]
Lifetime trauma exposure [Count of Participants; unit: Participants]
  Combat exposure | 357 | 347 | 704
  Any sexual trauma | 166 | 163 | 329
  Physical assault | 386 | 408 | 794
  Disaster exposure | 391 | 385 | 776
  Serious accident | 385 | 389 | 774
  Life-threatening illness or injury | 154 | 163 | 317
  Other traumatic event | 371 | 354 | 725
PTSD disability [Count of Participants; unit: Participants] — Two participants in the PE group and two participants in the CPT group did not report their "PTSD Disability" status. Population: Two participants in the PE group and two participants in the CPT group did not report their "PTSD Disability" status.
  Participants
    Approved: number analyzed (Participants) | 453 | 459 | 912
    Approved | 186 | 202 | 388
    Pending: number analyzed (Participants) | 453 | 459 | 912
    Pending | 116 | 129 | 245
    Denied: number analyzed (Participants) | 453 | 459 | 912
    Denied | 26 | 19 | 45
    Never applied: number analyzed (Participants) | 453 | 459 | 912
    Never applied | 125 | 109 | 234
Receiving psychotherapy [Count of Participants; unit: Participants] | 95 | 98 | 193
Taking psychotropic medication [Count of Participants; unit: Participants] | 303 | 317 | 620
Any current comorbid psychiatric disorder [Count of Participants; unit: Participants] | 343 | 371 | 714
Any current comorbid psychiatric disorder [Count of Participants; unit: Participants]
  Mood disorder | 309 | 332 | 641
  Anxiety disorder | 139 | 166 | 305
  Substance use disorders | 32 | 40 | 72
  Obsessive compulsive disorder | 19 | 29 | 48
Any lifetime comorbid psychiatric disorder [Count of Participants; unit: Participants] | 417 | 424 | 841
Any lifetime comorbid psychiatric disorder [Count of Participants; unit: Participants]
  Mood disorder | 398 | 400 | 798
  Anxiety disorder | 149 | 181 | 330
  Substance use disorders | 130 | 112 | 242
  Obsessive compulsive disorder | 24 | 36 | 60
Clinician Administered PTSD Scale-5 [Mean (Full Range); unit: score on a scale] — Possible range for CAPS-5 total score 0-80. Higher score indicates more severe PTSD.
  score on a scale | 39.9 [39.1 to 40.7] | 40.3 [39.5 to 41.1] | 40.1 [39.6 to 40.7]
Posttraumatic Diagnostic Scale [Mean (Full Range); unit: score on a scale] — Possible range for PDS-5 score 0-80. Higher PDS-5 Score indicates more severe PTSD Symptoms.
  score on a scale | 50.7 [49.5 to 52.0] | 50.5 [49.3 to 51.7] | 50.63 [49.8 to 51.5]
Beck Depression Inventory-II [Mean (Full Range); unit: score on a scale] — Possible range for BDI-II 0-63. Higher score indicates more severe depressive symptoms (0-13 minimal, 14-29 mild, 20-28 moderate, 29-63 severe).
  score on a scale | 30.3 [29.4 to 31.3] | 30.0 [29.0 to 30.9] | 30.2 [29.5 to 30.8]
Beck Depression Inventory-II Suicidality (BDI-II Item 9) [Count of Participants; unit: Participants] — Suicidality was coded by grouping "I have thoughts of killing myself, but I would not carry them out" "I would like to kill myself" and "I would kill myself if I had the chance" from item 9 of the BDI-II together as endorsing suicidality. Unit of measure is the #/% of participants who endorsed suicidality using this coding metric.
  Participants | 163 | 156 | 319
Spielberger Trait Anger Expression Inventory [Mean (Full Range); unit: score on a scale] — Subscale Ranges: State Anger 10-40, Trait Anger 10-40, Anger Expression 0-72. Higher score indicates more anger
  score on a scale
    State Anger | 17.8 [17.1 to 18.5] | 17.9 [17.3 to 18.6] | 17.9 [17.4 to 18.3]
    Trait Anger | 24.1 [23.5 to 24.8] | 24.2 [23.6 to 24.8] | 24.2 [23.7 to 24.6]
    Anger Expression | 37.3 [36.3 to 38.3] | 36.4 [35.5 to 37.4] | 36.9 [36.2 to 37.5]
Brief Addiction Monitor [Mean (Full Range); unit: score on a scale] — Range: 0-4 points. Higher score indicates worse outcome (i.e., more severe addiction)
  score on a scale | 0.8 [0.6 to 0.9] | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9]
Short Inventory of Problems-Revised [Mean (Full Range); unit: score on a scale] — Possible range for SIP-R 0-51. Higher score indicates more severe adverse consequences of substance use.
  score on a scale | 3.5 [2.7 to 4.3] | 3.3 [2.5 to 4.1] | 3.4 [2.9 to 4.0]
World Health Organization Disability Adjustment Scale-II [Mean (Full Range); unit: score on a scale] — Possible range for WHODAS-II 12-60. Higher score indicates more difficulty and disability due to health condition.
  score on a scale | 29.4 [28.6 to 30.3] | 29.7 [28.9 to 30.5] | 29.6 [29.0 to 30.1]
World Health Organization Quality of Life-BREF [Mean (Full Range); unit: score on a scale] — Possible range for WHOQOL-BREF 0-100, Physical Health 0-100, Psychological 0-100, Social Relationships 0-100, and Environment 0-100. Higher score indicates better satisfaction with life.
  score on a scale
    Physical Health | 44.4 [43.4 to 45.3] | 43.7 [42.7 to 44.7] | 44.1 [43.4 to 44.8]
    Psychological | 46.5 [45.2 to 47.8] | 46.4 [45.2 to 47.7] | 46.5 [45.6 to 47.4]
    Social Relationships | 41.3 [39.4 to 43.3] | 40.6 [38.7 to 42.5] | 41.0 [39.6 to 42.3]
    Environment | 58.2 [56.6 to 59.7] | 57.4 [55.9 to 59.0] | 57.8 [56.7 to 58.9]
Number of patients preferring PE treatment at baseline [Count of Participants; unit: Participants] — Treatment preference was assessed at baseline (before any treatment was administered, and before randomization to treatment arm had occurred). This measure is reported as the number of patients who reported a preference for PE as opposed to CPT. All unreported patients reported a preference for CPT (i.e., "no preference" was not a response option and no patients declined to answer).
  Participants | 232 | 214 | 446

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptom Severity on the Clinician-Administered PTSD Scale (CAPS)
Description: The primary outcome is the change of CAPS-5 total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). We chose to use the average in the six months post-treatment in the definition of primary outcome (versus using a single post-treatment timepoint) because we anticipate that improvement established during the course of treatment will be sustained in the 6 months after treatment for both PE and CPT. Possible range for CAPS-5 total score 0-80. Higher score indicates more severe PTSD.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 24.3 [22.8 to 25.2] | 27.2 [25.5 to 28.9]
  3 Months | 26.4 [25.1 to 27.8] | 28.7 [27.2 to 30.2]
  6 Months | 24.8 [23.2 to 26.2] | 26.9 [25.4 to 28.4]
Statistical Analysis 1: Comparison: Behavioral: Prolonged Exposure (PE) vs Behavioral: Cognitive Processing Therapy (CPT); Overall Treatment Effect Response Odds Ratio (OR). Response is defined as greater than or equal to 10 point improvement in severity; Test type: Superiority; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.00 to 1.65] — Odds ratios were calculated with CPT as the reference group and reflect the overall main effect of treatment across all outcome assessments (post-treatment, 3-months, and 6-months)
Statistical Analysis 2: Comparison: Behavioral: Prolonged Exposure (PE) vs Behavioral: Cognitive Processing Therapy (CPT); Overall Treatment Effect Loss of Diagnosis Odds Ratio (OR). Loss of Diagnosis is defined as Response, plus no longer meeting DSM-5 symptom criteria and severity less than 25; Test type: Superiority; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.12 to 1.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Behavioral: Prolonged Exposure (PE) vs Behavioral: Cognitive Processing Therapy (CPT); Overall Treatment Effect Remission Odds Ratio (OR). Remission is defined as loss of diagnosis plus severity less than 12; Test type: Superiority; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.24 to 2.00] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Posttraumatic Diagnostic Scale (PDS-5)
Description: The PDS-5 is a 24-item self-report measure that assesses PTSD symptom severity in the last month according to DSM-5 criteria. The outcome is the change of PDS-5 total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for PDS-5 score 0-80. Higher PDS-5 Score indicates more severe PTSD Symptoms.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 33.5 [31.3 to 35.6] | 36.7 [34.7 to 38.7]
  3 Months | 34.5 [32.5 to 36.4] | 37.5 [35.6 to 39.4]
  6 Months | 33.6 [31.6 to 35.5] | 36.7 [34.8 to 38.7]

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: BDI-II is a brief, self-report inventory designed to measure the severity of depression symptomatology. The outcome is the change of BDI-II total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for BDI-II 0-63. Higher score indicates more severe depressive symptoms (0-13 minimal, 14-29 mild, 20-28 moderate, 29-63 severe).
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 22.0 [20.5 to 23.5] | 22.7 [21.3 to 24.1]
  3 Months | 22.2 [20.9 to 23.5] | 23.6 [22.3 to 24.9]
  6 Months | 21.9 [20.6 to 23.3] | 22.9 [21.5 to 24.2]

4. Secondary Outcome: Spielberger State Anger Inventory (STAXI)
Description: The STAXI is a commonly used measure of trait and state anxiety. The outcome is the change of STAI total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for STAXI 44-176. Higher score indicates greater intensity of anger.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 93.4 [91.4 to 95.4] | 94.6 [92.7 to 96.5]
  3 Months | 93.2 [91.2 to 95.3] | 94.7 [92.8 to 96.6]
  6 Months | 93.2 [91.1 to 95.4] | 94.5 [92.6 to 96.4]

5. Secondary Outcome: Short Inventory of Problems - Revised (SIP-R)
Description: The SIP-R assesses alcohol-related consequences. The outcome is the change of SIP-R total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for SIP-R 0-51. Higher score indicates more severe adverse consequences of substance use.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 2.61 [1.89 to 3.34] | 2.49 [1.76 to 3.23]
  3 Months | 2.42 [1.58 to 3.25] | 2.29 [1.60 to 2.97]
  6 Months | 3.09 [2.22 to 3.95] | 1.72 [0.93 to 2.51]

6. Secondary Outcome: Brief Addiction Monitor (BAM)
Description: The BAM measures an individual's health, alcohol, and drug use. The outcome is the change of BAM total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Range: 0-4 points. Higher score indicates worse outcome (i.e., more severe addiction).
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 0.88 [0.73 to 1.03] | 0.86 [0.69 to 1.02]
  3 Months | 1.0 [0.84 to 1.16] | 0.94 [0.78 to 1.1]
  6 Months | 0.96 [0.82 to 1.11] | 0.80 [0.64 to 0.97]

7. Secondary Outcome: World Health Organization Disability Assessment Schedule (WHO-DAS-II)
Description: The WHO-DAS-II is an assessment instrument for health and disability. The outcome is the change of WHO-DAS-II total score from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for WHODAS-II 12-60. Higher score indicates more difficulty and disability due to health condition.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Posttreatment | 28.6 [27.7 to 29.4] | 28.6 [27.8 to 29.4]
  3 Months | 28.0 [27.1 to 29.0] | 28.7 [27.7 to 29.7]
  6 Months | 28.5 [27.5 to 29.4] | 28.5 [27.4 to 29.5]

8. Secondary Outcome: World Health Organization Quality of Life (WHOQoL-BREF)
Description: The WHOQoL-BREF is a quality of life assessment. The outcome is the change of WHOQoL-BREF assessment sub-category (Physical Health, Psychological, Social Relationships, Environment) scores from baseline (pre-treatment) to the average in the six months post-treatment (measured at immediate post-treatment, 3 and 6 months follow-up visits). Possible range for WHOQOL-BREF 0-100, Physical Health 0-100, Psychological 0-100, Social Relationships 0-100, and Environment 0-100. Higher score indicates better satisfaction with life.
Time Frame: immediate post-treatment, 3 and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 455 | 461
score on a scale
  Physical Health - Posttreatment | 47.0 [44.5 to 49.5] | 48.6 [46.0 to 51.1]
  Physical Health - 3 Months | 47.0 [45.7 to 48.2] | 47.0 [45.8 to 48.2]
  Physical Health - 6 Months | 47.1 [45.8 to 48.4] | 46.9 [45.6 to 48.2]
  Psychological - Posttreatment | 49.0 [47.5 to 50.5] | 48.9 [47.3 to 50.5]
  Psychological - 3 Months | 49.1 [47.7 to 50.5] | 48.1 [46.7 to 49.4]
  Psychological - 6 Months | 49.5 [47.9 to 51.1] | 49.1 [47.6 to 50.7]
  Social Relationship - Posttreatment | 45.4 [43.1 to 47.8] | 43.9 [41.6 to 46.3]
  Social Relationship - 3 Months | 46.2 [43.6 to 48.8] | 44.1 [41.6 to 46.6]
  Social Relationship - 6 Months | 46.2 [43.8 to 48.6] | 45.5 [42.8 to 48.2]
  Environment - Posttreatment | 61.1 [59.3 to 62.9] | 59.5 [57.6 to 61.3]
  Environment - 3 Months | 61.5 [59.8 to 63.2] | 59.8 [58.2 to 61.4]
  Environment - 6 Months | 62.3 [60.5 to 64.1] | 60.9 [59.2 to 62.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 12 months
Description: Adverse Events (AEs) related to the study intervention were collected from consent through completion of or termination from the study (approx. 12 months if patient completed study according to protocol, shorter if patient terminated from study participation early, longer if patient needed more time to complete assessment or treatment). All Serious Adverse Events (SAEs), regardless of relatedness, were collected from consent through 30 days post completion or termination from the study.
Groups:
- Behavioral: Prolonged Exposure (PE): Prolonged Exposure (PE) is a manualized, 90-minute, 8-15 week treatment program based on emotional processing theory, which posits that anxiety disorders, including PTSD, reflect pathological fear structures in which emotional and cognitive associations among different elements do not accurately represent reality and renders the individual dysfunctional and distressed. PE is designed to correct erroneous connections in the targeted memory structure. PTSD sufferers typically experience two key pathological emotional response sets and related cognitions: "The world is an utterly dangerous place," and "I am completely incompetent and unable to cope with stress." In this study, the 12-session protocol will be followed, but participants improve more rapidly may finish in 10 sessions and those who improve more slowly may have up to 2 additional sessions to continue working on exposure.
- Behavioral: Cognitive Processing Therapy (CPT): Cognitive Processing Therapy (CPT) consists of cognitive therapy and a written trauma narrative. Patients are taught to challenge their beliefs through Socratic questioning and the use of daily worksheets. The initial focus is on beliefs such as denial and self-blame, and then shifts to overgeneralized beliefs about self and the world. Patients process their trauma directly by writing a narrative of their traumatic event(s) that they read to themselves and to therapists. The typical protocol consists of 12 1-hr sessions. In this study, the 12-session protocol will be followed, but participants who improve more rapidly may finish in 10 sessions and those who improve more slowly may receive up to 2 additional sessions to continue working on stuck points with challenging beliefs worksheets.
Arm/Group | Behavioral: Prolonged Exposure (PE) | Behavioral: Cognitive Processing Therapy (CPT)
All-Cause Mortality (participants affected / at risk) | 1/455 | 2/461
Serious Adverse Events (participants affected / at risk) | 55/455 | 63/461
Other Adverse Events (participants affected / at risk) | 42/455 | 65/461
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral: Prolonged Exposure (PE) (N=455) | Behavioral: Cognitive Processing Therapy (CPT) (N=461)
Suicide attempt (Psychiatric disorders) | 1 (2) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Accidental Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adverse Drug Reaction (General disorders) | 2 (2) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (2)
Alcohol Detoxification (Surgical and medical procedures) | 2 (5) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (4)
Aortic aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood Glucose Decreased (Investigations) | 0 (0) | 1 (2)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1)
Breast Enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Calcinosis (General disorders) | 0 (0) | 1 (2)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive Symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Drug Administration Error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug Detoxification (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug Interaction (General disorders) | 0 (0) | 1 (1)
Drug Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Eye Operation Complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (6)
Hernia (General disorders) | 0 (0) | 1 (4)
Hernia Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (5)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (2) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infected Bite (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (3) | 0 (0)
Knee Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Localized Infection (Infections and infestations) | 1 (2) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 4 (6)
Neck Surgery (Surgical and medical procedures) | 0 (0) | 1 (8)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 0 (0)
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (2) | 3 (3)
Panic Disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Pharyngeal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Physical Assault (Social circumstances) | 0 (0) | 1 (7)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post-Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 1 (4) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (5) | 3 (3)
Scar excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Snake Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Fusion Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 6 (10) | 12 (18)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (2)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (9) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Violence-related symptom (Psychiatric disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral: Prolonged Exposure (PE) (N=455) | Behavioral: Cognitive Processing Therapy (CPT) (N=461)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (3) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 2 (3)
Alcoholism (Psychiatric disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Burglary Victim (Social circumstances) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Crying (General disorders) | 0 (0) | 1 (2)
Death of Companion (Social circumstances) | 0 (0) | 2 (3)
Death of Relative (Social circumstances) | 2 (4) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 1 (1)
Drug Administration Error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug screen positive (Investigations) | 0 (0) | 1 (1)
Drug Use Disorder (Psychiatric disorders) | 1 (2) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Electric Shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emotional Distress (Psychiatric disorders) | 1 (1) | 1 (1)
Exaggerated startle response (Nervous system disorders) | 0 (0) | 1 (1)
Eye Swelling (Eye disorders) | 0 (0) | 1 (1)
Facial Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Flashback (Psychiatric disorders) | 1 (2) | 1 (1)
Hallucination, Auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Homeless (Social circumstances) | 0 (0) | 1 (1)
Homicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hypervigilance (Psychiatric disorders) | 1 (1) | 0 (0)
Impaired Driving Ability (Social circumstances) | 0 (0) | 1 (1)
Imprisonment (Social circumstances) | 2 (2) | 4 (5)
Intentional Self-Injury (Psychiatric disorders) | 0 (0) | 2 (2)
Intrusive Thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Legal Problem (Social circumstances) | 3 (3) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Loss of Employment (Social circumstances) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Marital Problem (Social circumstances) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 3 (4)
Pain (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Physical Assault (Social circumstances) | 2 (3) | 6 (9)
Post-traumatic Stress Disorder (Psychiatric disorders) | 5 (8) | 4 (4)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Shoplifting (Social circumstances) | 1 (1) | 0 (0)
Sick Relative (Social circumstances) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 2 (3)
Substance Use (Social circumstances) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 6 (8) | 12 (18)
Suicide of Relative (Social circumstances) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapy Cessation (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Violence-related symptom (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The presentation or publication of any data collected by investigators on participants entered into the VA cooperative study is under the control of the study's Executive Committee. No individual participating investigator is permitted to perform analyses or interpretations or to make public presentations or seek publication of any of the data other than under the auspices and approval of the Executive Committee.

DOCUMENTS (3):
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT01928732/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT01928732/SAP_001.pdf
  • Informed Consent Form (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT01928732/ICF_002.pdf